CLINICAL TRIAL: NCT03455699
Title: Follow-up of Patients Treated in VeClose Study (Five Years)
Brief Title: VeClose Five Year Follow-Up Extension Study
Status: Completed | Type: Observational
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1011
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Great Saphenous Vein (GSV) With Venous Reflux Disease
Keywords: GSV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Experimental: VenaSeal SCS: Endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). The VA is dispensed in small amounts with each pull of the trigger equaling 0.10 cc. Subjects were randomized in a 1:1 ratio to either VenaSeal SCS or to RFA at the time of enrollment into the VeClose study (NCT01807585).
  Interventions: Device: VenaSeal SCS
- Active Comparator: RFA: Endovenous insertion of the ClosureFast radiofrequency ablation (RFA) catheter into a target site in diseased great saphenous veins (GSV). Heat is applied to the target vein using radiofrequency energy to ablate the target vein. Subjects were randomized in a 1:1 ratio to either VenaSeal SCS or to RFA at the time of enrollment into the VeClose study (NCT01807585).
  Interventions: Device: ClosureFast Radiofrequency Ablation (RFA)
- Experimental: Roll-in (VenaSeal SCS): Prior to initiation of the randomized cohort at each site for the VeClose study (NCT01807585), a non-randomized cohort of 2 subjects per site (roll-in phase) were enrolled and treated with VenaSeal SCS with endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). The VA is dispensed in small amounts with each pull of the trigger equaling 0.10 cc.
  Interventions: Device: Roll-In (VenaSeal SCS)

INTERVENTIONS:
Device: VenaSeal SCS — Non-tumescent, non-thermal, non-sclerosant procedure that uses a proprietary medical adhesive delivered endovenously to close the vein.
  Other Names: VenaSeal Sapheon Closure System; VSCS
  Groups: Experimental: VenaSeal SCS
Device: ClosureFast Radiofrequency Ablation (RFA) — Radiofrequency thermal ablation of the GSV using the Covidien ClosureFast system.
  Other Names: ClosureFast
  Groups: Active Comparator: RFA
Device: Roll-In (VenaSeal SCS) — Non-tumescent, non-thermal, non-sclerosant procedure that uses a proprietary medical adhesive delivered endovenously to close the vein.
  Other Names: VenaSeal Sapheon Closure System; VSCS; Roll-in
  Groups: Experimental: Roll-in (VenaSeal SCS)

SUMMARY:
The VeClose Five Year Follow-up Extension Study will seek to gain additional follow-up data from the patients enrolled in the VeClose study (NCT01807585).

DETAILED DESCRIPTION:
The VeClose Five Year Follow-up Extension Study will continue to assess the safety and efficacy of the VenaSeal Closure System for the long term effect on closure of the great saphenous vein by conducting a follow-up visit at five years post index procedure/enrollment in the VeClose study.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the VeClose study.
2. Able and willing to complete the required 5 year study visit including Duplex ultrasound exam.
3. Able and willing to provide written informed consent prior to study specific data collection.

Exclusion Criteria:

1. Withdrew consent from the VeClose study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects currently enrolled in both arms of the VeClose Study (NCT01807585) will be assessed for eligibility to enroll in the VeClose Five Year Follow-up Extension Study. All subjects must meet the inclusion criteria and must not meet the exclusion criteria. Assessment of eligibility is based on data available to the investigator at the time of subject enrollment. The subject will be considered to be enrolled in the VeClose Five Year Follow-up Extension Study after the informed consent is signed/dated and all of the study eligibility criteria have been met.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Complete Closure of the Target Vein at 5 years after index treatment in the VeClose study (NCT01807585). | 5 years
  Complete closure is defined as Doppler ultrasound examination showing closure along entire treated target vein segment with no discrete segments of patency exceeding 5cm.

SECONDARY OUTCOMES:
Venous Clinical Severity Score (VCSS) | 5 years
  Change in Venous Clinical Severity Score (VCSS) at 5 years as compared to baseline data from the VeClose study (NCT01807585). The VCSS is an Investigator assessment of the severity of venous reflux disease, assessing signs and symptoms such as pain, varicose veins, venous edema, skin pigmentation, induration and inflammation. The VCSS score is the sum of responses to 10 questions. Each question has a total possible of 3 points, which are then added for each question. The overall VCSS scores can therefore range from 0 (no venous disease) to 30 (severe venous disease). High scores indicate worse outcomes and "0" is the best possible outcome.
Aberdeen Varicose Vein Questionnaire (AVVQ) | 5 years
  Change in Aberdeen Varicose Vein Questionnaire (AVVQ) at 5 years as compared to baseline data from the VeClose study (NCT01807585). AVVQ is a disease-specific 13-item questionnaire used to assess the impact of varicose veins on the quality of life, such as pain caused by varicose veins, and need to take painkilling tablets for varicose veins as well as assessing the presence of signs/symptoms such as ankle swelling, purple discoloration and rash/eczema. The total score of AVVQ is the sum of all questions for each leg. Scores range from 0 (no disease) to 100 (maximal disease). High scores indicate worse outcomes and "0" is the best possible outcome.
Quality of Life survey (EQ-5D) | 5 years
  Change in Quality of Life survey (EQ-5D) at 5 years as compared to baseline data from the VeClose study (NCT01807585). EQ-5D is a short generic quality of life survey that is commonly used outside of the United States for health technology assessments. The "health state today" question provides an overall assessment along a 20-cm visual analog scale (VAS) with a range from 0 ("worst imaginable health state") to 100 ("best imaginable health state").
CEAP classification ("clinical, etiology, assessment and pathophysiology") | 5 years
  Standardized measure of the degree of venous insufficiency and secondary manifestations of venous disease as measured by the treating physician.
Satisfaction with Treatment | 5 years
  Satisfaction with Treatment assessment consists of a brief 2-question patient survey rating satisfaction with treatment provided and whether the subject would undergo the assigned treatment again. The number (percent) of subjects on each level of satisfaction are summarized (Very satisfied, Somewhat satisfied, Somewhat dissatisfied, Very dissatisfied). The number (percent) of subjects for the second satisfaction question, "would undergo treatment again" were also summarized by response (Definitely have again, Might have again, Not have again).
Adverse events (AE) related to the target GSV | 5 years
  AEs related to the GSV will be tabulated and reporting using the MedDRA dictionary, version 16.1.
Adjunctive procedures performed on the study limb | 5 years
  Details of adjunctive procedures performed on the study limb will be captured on Case Report Forms (CRFs)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Morrison, MD, Principal Investigator — Morrison Vein Institute
Locations (9):
- United States (9):
  - Morrison Vein Institute, Scottsdale, Arizona
  - GBK Cosmetic Laser Dermatology, San Diego, California
  - Radiology Imaging Associates (RIA), Greenwood Village, Colorado
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - MD Laser Skin & Vein Institute, Hunt Valley, Maryland
  - Vein Institute of Buffalo, North Tonawanda, New York
  - Inovia Vein Speciality Center, Bend, Oregon
  - Sentara Vascular Specialists, Virginia Beach, Virginia
  - Lake Washington Vascular, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morrison N, Gibson K, Vasquez M, Weiss R, Cher D, Madsen M, Jones A. VeClose trial 12-month outcomes of cyanoacrylate closure versus radiofrequency ablation for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2017 May;5(3):321-330. doi: 10.1016/j.jvsv.2016.12.005. Epub 2017 Mar 6. PMID 28411697
- [Background] Kolluri R, Gibson K, Cher D, Madsen M, Weiss R, Morrison N. Roll-in phase analysis of clinical study of cyanoacrylate closure for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2016 Oct;4(4):407-15. doi: 10.1016/j.jvsv.2016.06.017. Epub 2016 Aug 8. PMID 27638993
- [Derived] Morrison N, Gibson K, Vasquez M, Weiss R, Jones A. Five-year extension study of patients from a randomized clinical trial (VeClose) comparing cyanoacrylate closure versus radiofrequency ablation for the treatment of incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2020 Nov;8(6):978-989. doi: 10.1016/j.jvsv.2019.12.080. Epub 2020 Mar 20. PMID 32205125